CLINICAL TRIAL: NCT02954666
Title: Second Study on Cardio-neuromodulation in Humans
Acronym: CardNMH2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imelda Hospital, Bonheiden (Other)
Responsible Party: Principal Investigator, Philippe Debruyne, Principal investigator (PI), Head of Electrophysiology, Imelda Hospital, Bonheiden
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B689201629811
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Cardiac Disease; Syncope; Syncope, Vasovagal; Sick Sinus Syndrome
Keywords: cardio-neuromodulation; cardio-neuroablation; ablation; ganglionated plexi; anterior right ganglionated plexus; syncope
MeSH Terms: conditions — Heart Diseases; Syncope; Syncope, Vasovagal; Sick Sinus Syndrome | interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients with neurally mediated syncope (Experimental): Tailored radio-frequency ablation of the ARGP (CardNM).
  Interventions: Device: radio-frequency ablation
- Patients with sick sinus syndrome (Experimental): Tailored radio-frequency ablation of the ARGP (CardNM).
  Interventions: Device: radio-frequency ablation

INTERVENTIONS:
Device: radio-frequency ablation — Patients will undergo a tailored 'radio-frequency ablation' of the ARGP with the Smart Touch™ catheter or with the nMARQ™ catheter. Radiofrequency applications will be interrupted if no significant P-P interval shortening is observed after 30 seconds or if P-P interval is ≤ 550 ms during ablation.
  The ablation procedure is considered complete when one of the following conditions is fulfilled:
  P-P interval < 70% baseline procedural P-P interval after 5minute of waiting time; P-P interval < 600 ms after 5 minute of waiting time; 5 radiofrequency applications > 30 seconds have been delivered with the nMARQ™ catheter or 10 applications with the Smart Touch catheter.
  Other Names: cardio-neuromodulation, cardio-neuroablation, ARGP

SUMMARY:
Different approaches to cardio-neuroablation (CNA) to treat neurally mediated syncope, sinus node dysfunction, and functional atrioventricular block have been published. Investigators have developed a more limited and specific approach of CNA, called cardio-neuromodulation (CardNM). This treatment is based on a tailored vagolysis of the sinoatrial node through partial ablation of the anterior right ganglionated plexus (ARGP); it is also based on an innovative anatomic strategy. The feasibility of CardNM has already been tested in our center in a limited first study in humans (CardNMH1), with a favorable outcome for the patients involved. The results of CardNMH1 have been submitted for publication. The purpose of this second study of CardNM in humans (CardNMH2) is to collect more procedural and clinical data in well-defined patient groups.

DETAILED DESCRIPTION:
This is a phase II A prospective, interventional study. All patients will undergo CardNM. The study will involve eight different steps, from the screening procedure through study completion: screening, enrollment, pharmacological testing, group allocation, preprocedural assessment, procedure, follow-up, study completion.The dedicated study nurse and the PI are responsible for recording all data from the trial on the case report forms (CRFs) and completing the study database. A dedicated independent physician will be responsible for the safety monitoring. The PI will permit inspection of the trial files and the database by national or international official controlling scientific authorities, if required. The PI will review and monitor completed CRFs and the database at regular intervals throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

Candidates must meet all of the inclusion criteria required for inclusion in one of the two groups (summarized in Table 2). All of the patients need to have a positive P wave of > 0.5 mm in lead 2. Patients must have had ≥ 1 syncope during the 6 months preceding enrollment and ≥ 2 syncopes in their lifetime except if the last syncope was complicated by an injury or an accident, in which case further waiting for CardNM may be less desirable. Patients < 18 years must have least 3 syncopes with an interval exceeding 1 month unless 1 syncope was complicated by an injury or an accident.

If a significant rate drop (> 15%) is noted during head-up tilt test (HUT), either isolated or combined with vasoplegia, and associated with syncope or severe presyncope, patients will be eligible for inclusion in group A. If the HUT is negative and a pause > 3 seconds has been documented, patients will be assigned to group B. If both conditions are present, patients will be eligible for inclusion in either group but will be preferentially assigned to group A.

Exclusion Criteria:

Candidates will be excluded if ANY of the following criteria apply (detailed in Table 3):

* < 14 years of age;
* Inability to provide consent;
* Chronotropic negative medications (excepted in patients with a previous history of atrial fibrillation);
* 4 g amiodarone intake during the 2 months preceding enrollment;
* Alternating right bundle branch block (RBBB) and left bundle branch block (LBBB), HV interval > 70 ms;
* LBBB, bifascicular block (RBBB + left anterior hemiblock [LAHB], RBBB + left posterior hemiblock [LPHB]);
* PR interval permanently > 240 ms;
* Permanent AF, PAF or electrical cardioversion during the last 6 months;
* Valvular or subvalvular aortic stenosis, mitral stenosis;
* Any unstable medical condition, life expectancy < 12 months;
* Syncopes due a non-cardiac disease (excepted NMS) or advanced neuropathy;
* Current pregnancy;
* glaucoma.

Patients with transient atrioventricular conduction disturbances and normal atrioventricular conduction during an exercise test and normal QRS complexes are eligible for this study.

Patients with a high risk of bleeding are eligible, but clopidogrel (75 mg daily, 1 month of treatment) will then be preferred to oral anticoagulants.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
freedom from syncope | 12 months
freedom from serious adverse event | 7 days

SECONDARY OUTCOMES:
freedom from pre syncope | 12 months

OTHER OUTCOMES:
quantification of the vagolysis of the sinus node | procedure, 1,3,6,12 months
  The quantification of vagolysis of the sinus node obtained during CardNM will be evaluated by automatic P-P interval measurements during procedure, by ECG derived and standardized P-P interval measurements and by automatical quantification of P-P interval histograms on Holter registrations before procedure and during FU.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Debruyne, MD, Principal Investigator — Imeldahospital
Locations (1):
- Imeldaziekenhuis, Bonheiden, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debruyne P. "Cardio-Neuromodulation" With a Multielectrode Irrigated Catheter: A Potential New Approach for Patients With Cardio-Inhibitory Syncope. J Cardiovasc Electrophysiol. 2016 Sep;27(9):1110-3. doi: 10.1111/jce.13031. Epub 2016 Aug 1. PMID 27307200
- [Derived] Debruyne P, Rossenbacker T, Janssens L, Collienne C, Ector J, Haemers P, le Polain de Waroux JB, Bazelmans C, Boussy T, Wijns W. Durable Physiological Changes and Decreased Syncope Burden 12 Months After Unifocal Right-Sided Ablation Under Computed Tomographic Guidance in Patients With Neurally Mediated Syncope or Functional Sinus Node Dysfunction. Circ Arrhythm Electrophysiol. 2021 Jun;14(6):e009747. doi: 10.1161/CIRCEP.120.009747. Epub 2021 May 17. PMID 33999698
- [Derived] Debruyne P, Rossenbacker T, Collienne C, Roosen J, Ector B, Janssens L, Charlier F, Vankelecom B, Dewilde W, Wijns W. Unifocal Right-Sided Ablation Treatment for Neurally Mediated Syncope and Functional Sinus Node Dysfunction Under Computed Tomographic Guidance. Circ Arrhythm Electrophysiol. 2018 Sep;11(9):e006604. doi: 10.1161/CIRCEP.118.006604. PMID 30354289